CLINICAL TRIAL: NCT02378142
Title: A Phase II Evaluation of Pazopanib in the Treatment of Recurrent or Persistent Leiomyosarcoma of the Uterus
Brief Title: Pazopanib for Treating Uterine Leiomyosarcoma
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Gynecologic Oncology Group (Network)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Organization: GOG Foundation (Network)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GOG-3006
Record Dates: First submitted 2015-02-17; First posted 2015-03-04 (Estimated); Last update posted 2015-11-18 (Estimated); Status verified 2015-11

CONDITIONS: Uterine Leiomyosarcoma
MeSH Terms: interventions — pazopanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm 1 (Experimental): Pazopanib 800mg oral daily
  Interventions: Drug: Pazopanib

INTERVENTIONS:
Drug: Pazopanib

SUMMARY:
The purpose of this study is to test any good and bad effects of the study drug pazopanib.

ELIGIBILITY:
Inclusion Criteria:

* Recurrent or persistent leiomyosarcoma of the uterus.
* measurable disease.
* Patients must have at least one "target lesion" to be used to assess response on this protocol as defined by RECIST version 1.1 (Section 8.1).
* Patients must not be eligible for a higher priority GOG protocol, if one exists. In general, this would refer to any active GOG Phase III protocol.
* GOG Performance Status of 0, 1, or 2.
* Patients should be free of active infection requiring antibiotics (with the exception of uncomplicated UTI).
* Any hormonal therapy directed at the malignant tumor must be discontinued at least one week prior to registration. Hormonal therapy will not count as a prior regimen (either cytotoxic or non-cytotoxic).
* Any other prior therapy directed at the malignant tumor, including chemotherapy and immunologic agents, must be discontinued at least three weeks prior to registration.
* Any prior radiation therapy must be completed at least 2 weeks prior to registration.
* At least 4 weeks must have elapsed since the patient underwent any major surgery (for example, hysterectomy, resection of a metastatic nodule); placement of a central venous catheter is considered minor, not major and thus time from a minor procedure until treatment on study may be shorter than 4 weeks.
* Patients must have had at least one prior chemotherapeutic regimen for management of leiomyosarcoma.
* Patients may have had one additional chemotherapeutic regimen for management of leiomyosarcoma, for a total of two prior lines of therapy.
* Patients must have NOT received any non-cytotoxic (biologic or targeted) agents as part of their primary treatment or for management of recurrent or persistent disease. (Patients who were previously treated on GOG 0250, a randomized trial of gemcitabine-docetaxel plus bevacizumab or placebo, are eligible, provided that the patient is known to have been treated on the placebo-containing arm and did not receive prior bevacizumab)
* Absolute neutrophil count (ANC) greater than or equal to 1,500/mcl (1.5 x 109/L). Platelets greater than or equal to 100,000/mcl (100 x 109/L). Hemoglobin greater than or equal to 9 g/dL. Patients may not have had blood transfusion or platelet transfusion within 7 days of screening assessment.
* Creatinine less than or equal to 1.5 mg/dL (133 umol/L) or, if >1.5 mg/dl, then calculated creatinine clearance must be greater than or equal to 30 mL/min.
* Hepatic function:

  * Bilirubin less than or equal to 1.5 x ULN (subjects with Gilbert's syndrome and elevations of indirect bilirubin only are eligible).
  * AST and ALT less than or equal to 2.5 x ULN and alkaline phosphatase less than or equal to 2.5 x ULN.
  * Subjects who have BOTH bilirubin greater than ULN and AST/ALT greater than ULN are not eligible. (Specifically, if bilirubin is greater than 1 x ULN but less than or equal to 1.5 x ULN, THEN the AST and ALT must be less than or equal to ULN for patient to be eligible. If AST and /or ALT are greater than 1 x ULN but less than or equal to 2.5 x ULN, THEN the bilirubin must be less than or equal to ULN for patient to be eligible.)
* Urine Protein/ Creatinine Ratio (UPCR) must be less than 1 (or urinary protein less than 1 g/24 hours). -Blood coagulation parameters: PT such that international normalized ratio (INR) is less than or equal to 1.2 x ULN (Patients on anticoagulant therapy are eligible if their INR is stable, and in-range INR, usually between 2 and 3) and a PTT less than or equal to 1.2 x ULN.
* Patients must have signed an approved informed consent and authorization permitting release of personal health information.
* Patients who have met the pre-entry requirements specified in section 7.0.
* Patients of childbearing potential must have a negative serum pregnancy test prior to the study entry and be practicing an effective form of contraception.
* Patients must be 18 years or older.
* Patients must be capable of taking and absorbing oral medications.
* Any concomitant medications that are associated with a risk of QTc prolongation and/or Torsades de Pointes should be discontinued or replaced with drugs that do not carry these risks, if possible. Patients who must take medication with a risk of possible risk of Torsades de Pointes should be watched carefully for symptoms of QTc prolongation, such as syncope. See Appendix III for a list of concomitant medications associated with QTc and Torsades de Pointes.

Patients with personal or family history of congenital long QTc syndrome are NOT eligible.

* CYP3A4 Inhibitors: Strong inhibitors of CYP3A4 are prohibited. Grapefruit juice is also an inhibitor of CYP450 and should not be taken with pazopanib.
* CYP3A4 Inducers: Strong inducers of CYP3A4 are prohibited.
* CYP Substrates: Concomitant use of agents with narrow therapeutic windows that are metabolized by CYP3A4, CYP2D6, or CYP2C8 is not recommended.

Exclusion Criteria:

* Prior therapy with pazopanib.
* Patients with other invasive malignancies, with the exception of non-melanoma skin cancer, and other specific malignancies as noted in Sections 3.23 and 3.24, are excluded if there is any evidence of other malignancy being present within the last three years. Patients are also excluded if their previous cancer treatment contraindicates this protocol therapy.
* Patients who have received prior radiotherapy to any portion of the abdominal cavity or pelvis OTHER THAN for the treatment of uterine leiomyosarcoma within the last three years are excluded. Prior radiation for localized cancer of the breast, head and neck, or skin is permitted, provided that it was completed more than three years prior to registration, and the patient remains free of recurrent or metastatic disease.
* Patients who have received prior chemotherapy for any abdominal or pelvic tumor OTHER THAN for the treatment of uterine leiomyosarcoma within the last three years are excluded. Patients may have received prior adjuvant chemotherapy for localized breast cancer, provided that it was completed more than three years prior to registration, and that the patient remains free of recurrent or metastatic disease.
* Patient has been treated with an investigational agent or device within 30 days of entering the study.
* Patient is known to have history of active Hepatitis B or C.
* Patients with clinically significant cardiovascular disease. This includes:
* Patients must have blood pressure (BP) no greater than 140 mmHg (systolic) and 90 mmHg (diastolic) for eligibility. (Note: initiation of antihypertensive medications is permitted prior to study entry. At least 24 hours must have elapsed between antihypertensive medication initiation and BP measurement. At that time the BP should be measured 3 times, approximately 2 minutes apart, the 3 values should be averaged. This average or mean BP must be less than 140/90 mmHg.
* Myocardial infarction or unstable angina or cardiac angioplasty or cardiac stenting or coronary artery bypass graft surgery or symptomatic peripheral vascular disease within 6 months of the first date of pazopanib therapy.
* New York Heart Association (NYHA) Class II or greater congestive heart failure (Appendix II).
* Women who have received prior anthracycline (e.g., doxorubicin and/or liposomal doxorubicin) and who have an ejection fraction less than the institutional lower limit of normal will be excluded from the study. Patients with a prior life time exposure to doxorubicin (or liposomal doxorubicin) of greater than 300 mg/m2 are NOT eligible.
* CTCAE grade 2 or greater peripheral vascular disease.
* History of cerebrovascular accident (CVA, stroke), transient ischemic attack (TIA) or subarachnoid hemorrhage within six months of the first date of pazopanib therapy.
* Women with a baseline QTc >480 milliseconds.
* History of cerebrovascular accident, including transient ischemic attack, or pulmonary embolism, within the past 6 months. (Note: subjects with recent DVT only (no PE) who have been treated with therapeutic anticoagulation for at least six weeks are eligible).
* A patient with arterial thrombosis within 6 months prior to enrollment.
* Patients with history or evidence upon physical examination of CNS disease, including primary brain tumor, seizures not controlled with standard medical therapy or any brain metastases.
* Active bleeding or pathologic conditions that carry high risk of bleeding, such as known bleeding disorder, coagulopathy, or tumor involving major vessels.
* Serious, non-healing wound, ulcer, or bone fracture. This includes history of abdominal fistula, gastrointestinal perforation or intra-abdominal abscess within 28 days prior to the first date of pazopanib therapy. Patients with underlying lesions that caused the fistula or perforation in the past that have not been corrected.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to pazopanib.
* HIV-positive subjects on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with pazopanib. In addition, these subjects are at increased risk of lethal infections when treated with marrow-suppressive therapy. Appropriate studies will be undertaken in subjects receiving combination antiretroviral therapy when indicated.
* Patients who are pregnant or nursing. Patients who are lactating should discontinue nursing prior to the first dose of study drug and should refrain from nursing throughout the treatment period and for 14 days following the last dose of study drug.
* Patients with any condition that may increase the risk of gastrointestinal bleeding or gastrointestinal perforation, including but not limited to:

  * active peptic ulcer disease
  * known gastrointestinal intraluminal metastatic lesions with risk of bleeding (gastrointestinal serosa metastatic lesion are permitted)
  * inflammatory bowel disease (e.g., ulcerative colitis, Crohn's disease) or other gastrointestinal conditions with increased risk of perforation
  * history of abdominal fistula, gastrointestinal perforation, or intraabdominal abscess within 28 days prior to beginning study treatment
* History of hemoptysis in excess of 2.5 mL (1/2 teaspoon ) within 8 weeks prior to first dose of pazopanib.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection or psychiatric illness/social situations that would limit compliance with study requirements.
* Major surgery or trauma within 28 days prior to first dose of pazopanib. (procedures such as catheter placement or central venous access device placement are not considered major surgery)
* Patients with known endobronchial lesions and/or lesions infiltrating major pulmonary vessels that increase the risk of pulmonary hemorrhage. (Note, the presence of tumor that is touching but not infiltrating is acceptable; large protruding endobronchial lesion in the main or lobar bronchi are excluded; lesion extensively infiltrating the main or lobar bronchi are excluded)
* Patients who are unwilling or unable to discontinue use of prohibited medications for at least 14 days prior to the first dose of study drug and for the duration of the study (see APPENDIX III regarding concomitant medications for the section titled "prohibited medications").

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-03; Primary Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Event free survival | 6 months
  To estimate the proportion of patients with persistent or recurrent uterine leiomyosarcoma, who survive event-free for at least 6 months (EFS > 6 months; events associated with the endpoint are death, disease progression, or beginning a subsequent therapy) and the proportion of patients who have objective tumor response (complete or partial), treated with pazopanib.
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | Every 4 weeks
  To determine the nature and degree of toxicity of pazopanib in this cohort of patients

SECONDARY OUTCOMES:
Progression-free survival | Every 3 months from time from study entry to time of progression or death, whichever occurs first, assessed up to 5 years
  To estimate progression-free survival in patients with recurrent or persistent leiomyosarcoma of the uterus
Event-free survival | Every 3 months from time of study entry totime of progression or death, whichever occurs first, assessed up to 5 years
  To estimate event-free survival in patients with recurrent or persistent leiomyosarcoma of the uterus
Overall survival | Every 3 months from time of study entry totime of progression or death, whichever occurs first, assessed up to 5 years
  To estimate overall survival in patients with recurrent or persistent leiomyosarcoma of the uterus

CONTACTS AND LOCATIONS:
Overall Officials: Martee Hensley, MD, Study Chair — MSKCC